CLINICAL TRIAL: NCT01191827
Title: fMRI Cholinergic Mechanisms in Schizophrenia
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: MHBB-011-07F; NCT00692679 (obsolete NCT alias)
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- risperidone
- clozapine: Patients with schizophrenia treated with clozapine

SUMMARY:
This study aims to determine how clozapine treatment improves neuronal measures of sensory gating in subjects with schizophrenia.

DETAILED DESCRIPTION:
This study will use functional magnetic resonance imaging (fMRI) to study patients treated with risperidone, a commonly used neuroleptic that does not improves sensory gating, to those treated with clozapine to determine which brain areas are involved in clozapine's normalization of sensory gating in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* age 18-60 yrs

Exclusion Criteria:

* claustrophobia
* weight > 250 lbs
* metal in body other than dental fillings

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects with schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason R. Tregellas, PhD, Principal Investigator — VA Eastern Colorado Health Care System, Denver
Locations (1):
- VA Eastern Colorado Health Care System, Denver, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone: Patients with schizophrenia treated with risperidone
Period: Overall Study
Arm/Group | Risperidone | Clozapine
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Individuals with schizophrenia.
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone | Clozapine | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (10.9) | 34.0 (8.5) | 34.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Neuronal Response During Sensory Gating
Description: Neuronal response (blood oxygenation level dependent functional magnetic resonance imaging signal, relative to the global mean) during sensory gating. Sensory gating is defined as the process of filtering out unnecessary environmental stimuli.
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: % BOLD signal
Arm/Group | Risperidone | Clozapine
Number analyzed (Participants) | 20 | 20
% BOLD signal | .12 (.1) | .11 (.1)

ADVERSE EVENTS:
Description: Serious/non-serious adverse events related to group membership were not assessed for this observational study.
Arm/Group | Risperidone | Clozapine
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes